CLINICAL TRIAL: NCT06465602
Title: Nicotinamide Supplementation Improves Physical Performance in Older Adults at Risk of Falls: a Pilot Randomized Clinical Trial
Brief Title: Nicotinamide Supplementation Improves Physical Performance in Older Adults at Risk of Falls
Acronym: NICE-FIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Centro FONDAP de Gerociencia, Salud mental y Metabolismo (GERO) (Unknown); Center for Advanced Clinical Research (CICA ) - University of Chile (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FONDAP 15150012 GERO
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-04

CONDITIONS: Frailty; Fall; Frailty Syndrome; Falls
Keywords: nicotinamide; Nicotinamide supplementation; motor rehabilitation; rehabilitation; exercise; falls; older adults; accidental falls; frail older adults; dietary supplementation
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: Pilot randomized clinical trial, block allocation, double-blind
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be assigned to either Nicotinamide or placebo through block allocation. One researcher will be responsible for patient recruitment via telephone and obtaining informed consent. Another researcher will perform patient randomization and drug dispensing. Physiotherapists conducting both the initial and final physical assessments and those conducting rehabilitation sessions will be blinded to the patient's assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide supplementation group (Experimental): At the beginning and end of the study, blood samples will be taken for the measurement of IL-6, CCL2, TNF-alpha, and NFL, and participants will be assessed using the Short Physical Performance Battery (SPPB), quadriceps dynamometry (LY-D Lynx Dynamo), quadriceps oxygen saturation (with NIRS), and posturography to determine the center of pressure (COP) area with the HUR BTG4 posturography system, and SmartBalance® software. Subjects will receive 1.5 grams per day of nicotinamide, orally, for 30 days. During this period, they will undergo a home-based physical training program guided by a physiotherapist. The sessions will be 50 minutes long (10 minutes warm-up, 30 minutes strength and balance training, and 10 minutes flexibility), twice a week.
  Interventions: Drug: Nicotinamide
- Placebo group (Placebo Comparator): Same physical evaluation and blood sampling as the experimental group. The subjects will receive 1.5 grams per day of placebo (talc, the medium in which nicotinamide is prepared), orally, for 30 days. The bottle and the capsules will be of the same physical characteristics (shape, color, and flavor) in both groups. During that period, patients will assess patient adherence and possible adverse effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide — The subjects will receive 1.5 grams per day of Nicotinamide, orally, for 30 days.
  Other Names: Niacinamide
  Arms: Nicotinamide supplementation group
Drug: Placebo — The subjects will receive 1.5 grams per day of placebo, orally, for 30 days.
  Arms: Placebo group

SUMMARY:
Falls are unplanned events resulting in contact with a lower surface. They are common in older adults, affecting one in three individuals over 65 years old. They have serious consequences, ranging from physical injuries (fractures, traumatic brain injury) to psychological repercussions. Physical training focused on muscle strength, balance, and gait has consistently been shown to prevent falls. However, there are significant challenges in its implementation, such as the need for trained personnel and long intervention times, which are associated with high costs. Therefore, developing strategies to improve the efficiency of physical training programs in older adults is mandatory. The reduced response to physical training in older adults compared to younger individuals is a well-documented phenomenon, reflecting physiological changes associated with aging.

Nicotinamide adenine dinucleotide (NAD+) is an essential coenzyme for cells, mediating energy metabolism and participating in crucial processes such as DNA repair, mitochondrial function, and cell death. As we age, NAD+ levels decrease in various tissues (including the brain and muscle), contributing to the development of aging phenotypes and associated pathologies. Preclinical evidence suggests that increasing NAD+ levels reduces the appearance of aging phenotypes. During physical activity, cellular metabolic pathways that increase the demand for NAD+ to support energy production in mitochondria are activated. This increase in demand is associated with the upregulation of key enzymes involved in NAD+ degradation promoted by exercise. Considering the decrease in cellular levels of this coenzyme associated with aging, it can be hypothesized that NAD+ deficiency may play a significant role in the reduced response of older adults to training programs. Nicotinamide, a water-soluble form of vitamin B3 currently considered a nutritional supplement, is a fundamental precursor for NAD+ synthesis, capable of raising cellular levels of it. It has already been used in clinical practice in the treatment of certain endocrinological and dermatological conditions. This study aims to determine through a randomized clinical trial whether nicotinamide supplementation improves physical performance in older adults at risk of falls undergoing a physical training program.

DETAILED DESCRIPTION:
To test the hypothesis, a randomized pilot clinical trial will be conducted using block allocation, double-blind (patient and evaluator), designed according to the SPIRIT guidelines for drafting a trial protocol. This study involves the implementation of guided home-based physical training by a physiotherapist (2 sessions per week for 4 weeks) combined with supplementation with nicotinamide (1.5 g/day) or placebo depending on the assigned group. Improvement in physical performance will be evaluated using the Short Physical Performance Battery (SPPB), handgrip strength test, quadriceps dynamometry, posturography, and near-infrared spectroscopy (NIRS) of the quadriceps. The RedCap software will be used for randomization and data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Living in the community
* Increased risk of falls, defined as:
* More than two falls in the last 12 months or
* Altered balance test (unable to maintain unipedal stance > 5 seconds) or
* SPPB score less than 10 points

Exclusion Criteria:

* Known Muscle Disease (dystrophy, myopathy, or similar)
* Motor sequelae of stroke
* Joint pathology with severe pain preventing strength exercises
* Cognitive impairment that renders the informed consent process impossible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement in physical performance | Four weeks
  Assess the change in total Short Physical Performance Battery (SPPB) performance from baseline to post-4 weeks

SECONDARY OUTCOMES:
Posturography | Four weeks
  Change Center of pressure (COP) between baseline and post-training in posturography
Dynamometry | Four weeks
  Change in dynamometry performance between baseline and post-training
Quadriceps saturation | Four weeks
  Change in quadriceps saturation after a 5-squat test
Adherence to medication | Four weeks
  Nicotinamide/placebo usage via self-report survey
Adverse effects | Four weeks
  Assessment of adverse effects using a standardized evaluation guideline.
Plasma sample analysis | Four weeks
  Nicotinamide leves, Interleukin-13 (IL-13), Interleukin-1(IL-1), Interleukin-6 (IL-6), mixed lineage kinase domain-like (MLKL), receptor interacting protein kinase 3 (RIPK3) and chemokine C-C ligand 2 (CCL-2)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe H Salech Morales, MD-PhD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrose AF, Paul G, Hausdorff JM. Risk factors for falls among older adults: a review of the literature. Maturitas. 2013 May;75(1):51-61. doi: 10.1016/j.maturitas.2013.02.009. Epub 2013 Mar 22. PMID 23523272
- [Background] Tsao YL, Hsu CC, Chen KT. Blunt Traumatic Retropharyngeal Hematoma with Respiratory Symptoms: A Systematic Review of Reported Cases. Emerg Med Int. 2021 Oct 7;2021:5158403. doi: 10.1155/2021/5158403. eCollection 2021. PMID 34659833
- [Background] Hayes WC, Myers ER, Morris JN, Gerhart TN, Yett HS, Lipsitz LA. Impact near the hip dominates fracture risk in elderly nursing home residents who fall. Calcif Tissue Int. 1993 Mar;52(3):192-8. doi: 10.1007/BF00298717. PMID 8481831
- [Background] Florence CS, Bergen G, Atherly A, Burns E, Stevens J, Drake C. Medical Costs of Fatal and Nonfatal Falls in Older Adults. J Am Geriatr Soc. 2018 Apr;66(4):693-698. doi: 10.1111/jgs.15304. Epub 2018 Mar 7. PMID 29512120
- [Background] Loureiro V, Gomes M, Loureiro N, Aibar-Almazan A, Hita-Contreras F. Multifactorial Programs for Healthy Older Adults to Reduce Falls and Improve Physical Performance: Systematic Review. Int J Environ Res Public Health. 2021 Oct 15;18(20):10842. doi: 10.3390/ijerph182010842. PMID 34682586
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Rodrigues F, Domingos C, Monteiro D, Morouco P. A Review on Aging, Sarcopenia, Falls, and Resistance Training in Community-Dwelling Older Adults. Int J Environ Res Public Health. 2022 Jan 13;19(2):874. doi: 10.3390/ijerph19020874. PMID 35055695
- [Background] Sun M, Min L, Xu N, Huang L, Li X. The Effect of Exercise Intervention on Reducing the Fall Risk in Older Adults: A Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2021 Nov 29;18(23):12562. doi: 10.3390/ijerph182312562. PMID 34886293
- [Background] Sherrington C, Fairhall NJ, Wallbank GK, Tiedemann A, Michaleff ZA, Howard K, Clemson L, Hopewell S, Lamb SE. Exercise for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD012424. doi: 10.1002/14651858.CD012424.pub2. PMID 30703272
- [Background] Chen Y, Zhang Y, Guo Z, Bao D, Zhou J. Comparison between the effects of exergame intervention and traditional physical training on improving balance and fall prevention in healthy older adults: a systematic review and meta-analysis. J Neuroeng Rehabil. 2021 Nov 24;18(1):164. doi: 10.1186/s12984-021-00917-0. PMID 34819097
- [Background] Adjetey C, Karnon B, Falck RS, Balasubramaniam H, Buschert K, Davis JC. Cost-effectiveness of exercise versus multimodal interventions that include exercise to prevent falls among community-dwelling older adults: A systematic review and meta-analysis. Maturitas. 2023 Mar;169:16-31. doi: 10.1016/j.maturitas.2022.12.003. Epub 2023 Jan 9. PMID 36630860
- [Background] Angulo J, El Assar M, Alvarez-Bustos A, Rodriguez-Manas L. Physical activity and exercise: Strategies to manage frailty. Redox Biol. 2020 Aug;35:101513. doi: 10.1016/j.redox.2020.101513. Epub 2020 Mar 20. PMID 32234291
- [Background] Alvarez C, Ramirez-Campillo R, Ramirez-Velez R, Izquierdo M. Effects and prevalence of nonresponders after 12 weeks of high-intensity interval or resistance training in women with insulin resistance: a randomized trial. J Appl Physiol (1985). 2017 Apr 1;122(4):985-996. doi: 10.1152/japplphysiol.01037.2016. Epub 2017 Feb 2. PMID 28153946
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349
- [Background] Covarrubias AJ, Perrone R, Grozio A, Verdin E. NAD+ metabolism and its roles in cellular processes during ageing. Nat Rev Mol Cell Biol. 2021 Feb;22(2):119-141. doi: 10.1038/s41580-020-00313-x. Epub 2020 Dec 22. PMID 33353981
- [Background] Ji LL, Yeo D. Maintenance of NAD+ Homeostasis in Skeletal Muscle during Aging and Exercise. Cells. 2022 Feb 17;11(4):710. doi: 10.3390/cells11040710. PMID 35203360
- [Background] Hwang ES, Song SB. Possible Adverse Effects of High-Dose Nicotinamide: Mechanisms and Safety Assessment. Biomolecules. 2020 Apr 29;10(5):687. doi: 10.3390/biom10050687. PMID 32365524
- [Background] Knip M, Douek IF, Moore WP, Gillmor HA, McLean AE, Bingley PJ, Gale EA; European Nicotinamide Diabetes Intervention Trial Group. Safety of high-dose nicotinamide: a review. Diabetologia. 2000 Nov;43(11):1337-45. doi: 10.1007/s001250051536. PMID 11126400
- [Background] Preyat N, Rossi M, Kers J, Chen L, Bertin J, Gough PJ, Le Moine A, Rongvaux A, Van Gool F, Leo O. Intracellular nicotinamide adenine dinucleotide promotes TNF-induced necroptosis in a sirtuin-dependent manner. Cell Death Differ. 2016 Jan;23(1):29-40. doi: 10.1038/cdd.2015.60. Epub 2015 May 22. PMID 26001219